CLINICAL TRIAL: NCT00099086
Title: Phase I Trial of Concurrent Taxotere With Radiation Therapy and Hormonal Therapy For Clinically Localized High Risk Prostate Cancer
Brief Title: Docetaxel, Radiation Therapy, and Hormone Therapy in Treating Patients With Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100783; HR 11326 (Other: MUSC IRB)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Docetaxel; Gonadotropin-Releasing Hormone; Goserelin; Leuprolide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: Bicalutamide; Drug: docetaxel; Drug: GnRh analog; Radiation: radiotherapy

INTERVENTIONS:
Drug: Bicalutamide — Bicalutamide will be administered for approximately 28 months: prior to radiotherapy (2 months), during radiotherapy (2 months), and after radiotherapy (24 months)
  Other Names: Casodex
Drug: docetaxel — Docetaxel will be administered weekly during radiotherapy. The docetaxel dose will be escalated as part of the study. Dose levels are: 10mg/m2; 15 mg/m2; 20 mg/m2 and 25 mg/m2
  Other Names: Taxotere
Drug: GnRh analog — A GnRH analog (goserelin acetate, leuprolide acetate) will be administered for approximately 28 months: prior to radiotherapy (2 months), during radiotherapy (2 months), and after radiotherapy (24 months)
  Bicalutamide will be administered for approximately 28 months: prior to radiotherapy (2 months), during radiotherapy (2 months), and after radiotherapy (24 months)
  Other Names: Zoladex; goserelin acetate; leuprolide acetate; Lupron
Radiation: radiotherapy — External beam photon radiotherapy utilizing 3-D-conformal or intensity modulated radiotherapy (IMRT) shall be used to deliver 77.4 4 Gy in 43 fractions of 1.8 Gy fractions.

SUMMARY:
This phase I trial is studying the side effects and best dose of docetaxel when given with radiation therapy and hormone therapy in patients with locally advanced prostate cancer.

DETAILED DESCRIPTION:
Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Docetaxel may also make tumor cells more sensitive to radiation therapy. Androgens can cause the growth of prostate cancer cells. Drugs, such as leuprolide, goserelin, or bicalutamide, may stop the adrenal glands from making androgens. Giving chemotherapy with radiation therapy and hormone therapy may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate with one of the prognostic factors specified in the protocol. No pelvic lymph node disease that would necessitate pelvic radiotherapy. No radiologic evidence of metastatic disease on bone scan or on CT scan or MRI of the abdomen or pelvis
2. No prior radiation therapy, chemotherapy, immunotherapy or alternative therapy for prostate cancer. Greater than 4 weeks since any major surgery.
3. Performance status 0-2
4. Must meet criteria for acceptable lab values as outlined in the protocol.
5. Peripheral neuropathy must be greater than or equal to 1
6. Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

1. No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with Polysorbate 80

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01-16 (Actual); Primary Completion 2011-01-20 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Taxotere with radiation therapy and hormonal therapy | 57 days
  To determine the MTD of Taxotere with radiation therapy and hormonal therapy in patients with high risk locally advanced adenocarcinoma of the prostate. The dose limiting toxicity (CLT) period for determining the MTD is 57 days.

CONTACTS AND LOCATIONS:
Overall Officials: David Marshall, MD, Principal Investigator — Medical University of South Carolina